CLINICAL TRIAL: NCT04969237
Title: Vitamine D in Post-COVID Patients
Acronym: VD-PCS
Status: Completed | Type: Observational
Sponsor: Klinikum Emden (Other)
Responsible Party: Principal Investigator, Jens Bräunlich, investigator, Klinikum Emden
Other Study IDs: 1
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Post COVID
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy subjects 2019: subjects with diseases not influencing vitamine D values without substitution nor post-COVID
  Interventions: Diagnostic Test: Vitamine D in blood samples
- healthy subjects 2020: subjects with diseases not influencing vitamine D values without substitution nor post-COVID
  Interventions: Diagnostic Test: Vitamine D in blood samples
- healthy subjects 2021: subjects with diseases not influencing vitamine D values without substitution nor post-COVID
  Interventions: Diagnostic Test: Vitamine D in blood samples
- post-COVID subjects 2021: subjects with diseases not influencing vitamine D values without substitution with diagnosed post-COVID syndrome
  Interventions: Diagnostic Test: Vitamine D in blood samples

INTERVENTIONS:
Diagnostic Test: Vitamine D in blood samples — vitamine D values

SUMMARY:
In this study routineously collected vitamine D values will compared to healthy cohorts from this year and previous years.

ELIGIBILITY:
Inclusion Criteria:

* patients with or without post-COVID-Syndrome

Exclusion Criteria:

* substitution of vitamine D
* diseases influencing vitamine D level

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy subjects and patients with post-COVID
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
vitamin D values between the groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Emden, Emden, Germany

IPD SHARING:
Plan to Share IPD: Undecided